CLINICAL TRIAL: NCT02521064
Title: The Role of Exclusive Enteral Nutrition in the Pediatric Inflammatory Bowel Disease Microbiome: a Pilot Study
Brief Title: Effects of Exclusive Enteral Nutrition on the Microbiome in Pediatric Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: McMaster Children's Hospital (Other)
Collaborators: Canadian Association of Gastroenterology (Industry)
Responsible Party: Principal Investigator, Lara Hart, Resident/fellow principal investigator, McMaster Children's Hospital
Other Study IDs: McmasterCH - 15-365
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; enteral nutrition; corticosteroids
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bl
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exclusive Enteral Nutrition (EEN): The patient will be admitted to hospital for placement of the nasogastric tube and commencement of exclusive enteral nutrition (EEN). Nutritional feeds will consist of a semi-elemental (whey-peptide based) formula that will make up all of the patient's daily caloric needs (120% of BMR). Feeds will slowly be titrated up to full volume and strength during the hospital stay. The patient will receive instructions how to decrease the number of hours of feeds once at home. The patient will be seen in clinic at two weeks and will receive a phone call from the dietician at 4 weeks to assess progress and symptom improvement. At 8 weeks, food will start to be reintroduced slowly, as per the dietician's instructions.
  Interventions: Dietary Supplement: Exclusive Enteral Nutrition (EEN)
- Prednisone: Patients who receive the prednisone intervention will follow the Division of Pediatric Gastroenterology and Nutrition protocol for corticosteroid induction therapy, with 2 weeks of high dose IV/PO prednisone (maximum 40mg/day) followed by a 6 week wean (approximately decreasing 5mg/day per week). The patient will receive a phone call from the nurse practitioner at two weeks and will be seen in clinic at 4 weeks to assess progress and symptom improvement.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Dietary Supplement: Exclusive Enteral Nutrition (EEN) — Patients will be treated with 8 weeks of Exclusive Enteral Nutrition (EEN). Patients will continue to receive usual medical care, and concurrent IBD treatments will be permitted.
  Other Names: Peptamen 1.5
  Groups: Exclusive Enteral Nutrition (EEN)
Drug: Prednisone — Patients will be treated with 8 weeks of prednisone (corticosteroid). Patients will continue to receive usual medical care, and concurrent IBD treatments will be permitted.
  Other Names: Corticosteroid
  Groups: Prednisone

SUMMARY:
Children with Crohn's disease can be effectively treated by remaining on a single-formula diet for 8 continuous weeks. This dietary therapy is known as "exclusive enteral nutrition" (EEN). It is just as effective as steroid treatment, which is what's traditionally used for the initial treatment of Crohn's disease. It is not clear why EEN is an effective treated. One possibility is that it changes the bacteria in our intestines, which allows the intestine to heal. It is also unclear whether EEN can be used to treat ulcerative colitis, a disease that is very similar to Crohn's disease. The purpose of our research project is to determine whether EEN can be used to treat ulcerative colitis, and understand how the intestinal bacteria changes while on EEN. Investigators will compare the results to patients who have either Crohn's disease or ulcerative colitis, and are receiving standard treatment for their disease (steroids). This is a pilot study, meaning that the goal of this study is to determine whether a larger study is feasible. Investigators will measure patient recruitment rates, whether patients are able to perform the treatment as requested, whether there are any safety concerns, and whether investigators are able to collect the bloodwork and stool samples without difficulty.

DETAILED DESCRIPTION:
Exclusive enteral nutrition (EEN) is an effective induction therapy in pediatric Crohn's disease (CD). Compared to corticosteroids, EEN has equivalent rates of clinical remission and significantly higher rates of mucosal healing and weight gain. There is a paucity of literature on the role of EEN in ulcerative colitis (UC). Some have postulated that colonic disease will not respond to EEN, yet two series found no difference in rates of clinical remission between small intestinal and colonic CD. The mechanisms underlying the effectiveness of enteral nutrition in colitis remain unclear. A microbiome-mediated pathogenesis is possible. Two studies have shown how EEN produces profound changes in microbial community structure within as little as 24 hours. These changes correlated with improved disease activity scores. Active inflammatory bowel disease also carries distinct microbial signatures. Baseline differences in taxonomy between IBD phenotypes may account for differences in EEN efficacy between CD and UC.

The purpose of the pilot study is to investigate if EEN can be used for induction of remission of ulcerative colitis, and compare its usage to a) corticosteroids for UC and b) EEN or corticosteroids for Crohn's disease. The goal is to eventually characterize the clinical, biochemical and microbial changes that occur with each. However, given that EEN is a challenging commitment, as a sole source of nutrition for 8 weeks, investigators first have to evaluate feasibility in terms of participant recruitment, compliance and safety of this treatment. Both EEN and corticosteroid treatment require proper compliance to be effective, which can be a significant burden for the patient and his/her family. Investigators will therefore also determine satisfaction with the induction therapies and effect on quality of life. Further, since frequent follow up is being requested, investigators need to assess recruitment and retention rates, as well as compliance with completing bloodwork and providing stool samples. Investigators hypothesize that these induction therapies will be both feasible and safe. However, it is anticipated that, while patients will be satisfied with the treatment, it may have a significant impact on quality of life during those 8 week.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-18 years old who have been diagnosed with IBD (confirmed by endoscopy, histology and radiography), and are followed by McMaster Children's Hospital's Division of Pediatric Gastroenterology and Nutrition.
* Patients requiring induction therapy
* Patients already taking 5-aminosalicylic acid (5-ASA) azathioprine, 6-mercaptopurine or anti-TNF (tissue necrosis factor) therapy (e.g. infliximab)

Exclusion Criteria:

* Patients who are in remission (on maintenance therapy).
* Patients who receive new medical therapies (e.g. antibiotics, probiotics) during the study period

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (<18yo) being followed and managed through the McMaster Children's Hospital's Division of Pediatric Gastroenterology. Patients are diagnosed with Crohn's Disease, Ulcerative Colitis, or Inflammatory Bowel Disease-Unclassified.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Feasibility: Participant recruitment rate | Entirety of study (1 year)
  Number of participants recruited per month
Feasibility: Participant retention rate | Entirety of study (1 year)
  Number of participants enrolled who did not complete the study
Feasibility: Participant compliance with intervention: treatment (EEN or corticosteroids) | Entirety of study (1 year)
  Number of participants who completed full treatment duration
Feasibility: Participant compliance with intervention: bloodwork, stool and urine sampling | Entirety of study (1 year)
  Number of blood, stool and urine sample collections per participant
Feasibility: Participant compliance with weekly interviews | Entirety of study (1 year)
  Number of weekly interviews completed per participant
  * Interviews discussing: a) disease assessment (Pediatric Ulcerative Colitis Activity Index [PUCAI]/Pediatric Crohn's Disease Activity Index [PCDAI] scores), and b) quality of life (health-related quality of life questionnaire)
Feasibility: Rate of adverse events in patients with ulcerative colitis receiving EEN | Entirety of study (1 year)
  Record of all adverse events

SECONDARY OUTCOMES:
Changes in microbiome (composite measure) | Entirety of study (1 year)
  Changes in microbial community structure in patients receiving EEN versus corticosteroid induction therapy. Multiple indices of alpha and beta diversity will comprise composite assessment of microbiome change.
Clinical remission (composite measure) | Entirety of study (1 year)
  Effects of EEN therapy on induction of clinical remission in pediatric UC versus CD. Composite assessment consisting of:
  1. 8 weeks: PUCAI Δ ≥20; PCDAI Δ ≥15, decrease in serum ESR, CRP, and fecal calprotectin
  2. 12 weeks: PUCAI <10; PCDAI <15, Normalization of serum ESR, CRP and fecal calprotectin)
Patient satisfaction and quality of life | Entirety of study (1 year)
  Patient satisfaction with the treatment (satisfaction validated questionnaire)
Patient quality of life | Entirety of study (1 year)
  Quality of life during induction therapy (quality of life validated questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Pai, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada